CLINICAL TRIAL: NCT06291077
Title: Comparison of the Effects of Belatacept and Anticalcineurins on Endothelial Function in Renal Transplant Patients <BELAFENDO>
Brief Title: Comparison of the Effects of Belatacept and Anticalcineurins on Endothelial Function in Renal Transplant Patients - <BELAFENDO>
Acronym: BELAFENDO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0391/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belatacept group (Experimental): Belatacept group
  Interventions: Drug: Belatacept
- anticalcineurin group (Active Comparator): anticalcineurin group
  Interventions: Drug: anticalcineurins

INTERVENTIONS:
Drug: Belatacept — Changing of anticalcineurins by Belatacept
  Arms: Belatacept group
Drug: anticalcineurins — Keeping of anticalcineurins
  Arms: anticalcineurin group

SUMMARY:
Kidney transplantation is the standard treatment for patients with end-stage renal failure.

However, anticalcineurin inhibitors, the most widely used immunosuppressants, are involved in the occurrence of cardiovascular events, a major cause of premature death in these patients. They play an important role in the occurrence of endothelial dysfunction and increased arterial stiffness by decreasing the synthesis of nitric oxide (NO), promoting intrarenal arterial vasoconstriction and stimulating the production of pro-inflammatory cytokines. leading to the development of hypertension and chronic graft dysfunction.

Belatacept, a more recently developed immunosuppressant and co-stimulation signal inhibitor, has shown an anti-rejection effect similar to cyclosporine with a better cardiovascular tolerance profile. Preliminary studies are contradictory on the influence of Belatacept on arterial stiffness. Furthermore, to date, no study has evaluated the impact of Belatacept on vasomotor endothelial function in humans, an indicator of NO bioavailability. The interest of this study is to demonstrate that patients taking Belatacept have an improvement in vascular function compared to patients taking anticalcineurins in order to consider an earlier change in immunosuppressive strategy in the event of vascular damage.

ELIGIBILITY:
Inclusion Criteria:

For the Belatacept group:

- Patients who have undergone a graft biopsy due to impaired renal function finding criteria for chronic toxicity of anticalcineurins leading to the introduction of Belatacept.

For the anticalcineurin group:

* Renal transplant patients treated with anticalcineurins for more than a year.
* Stable renal function (defined by a creatinine level in µmol/l stable for 3 months (variation +/-20%)

For both groups:

* Date of kidney transplant greater than 1 year
* Age between 18 and 75 years inclusive
* Patient having received clear information from one of the investigators, having read and understood the information letter and signed the consent form
* Women :

  * of childbearing age (defined by the CTFG as a fertile woman, after menarche and until menopause, except in cases of permanent sterility (including hysterectomy, bilateral salpingectomy or bilateral oophorectomy)

    * using effective contraception according to the WHO (combined hormonal contraception (containing estrogens and progestins), progestin-only contraception, intrauterine device (IUD), male or female condoms) for at least 4 weeks before inclusion and during the study And,
    * presenting a negative urine pregnancy test at inclusion;
  * menopausal: menopause according to the CTFG is defined as the absence of periods for 12 months without any other medical cause. An elevated follicle-stimulating hormone (FSH) level in the postmenopausal interval can be used to confirm a postmenopausal state in women who are not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* Patient benefiting from a social protection scheme

Exclusion Criteria:

* Stage 5 chronic renal failure (defined by a CKD-EPI GFR<15 ml/min/1.73m²)
* Dialysis patient
* History of myocardial infarction or stroke less than 6 months old
* Systolic heart failure requiring hospitalization in the 6 months preceding inclusion or known heart failure with an LVEF <30%
* BMI>35 kg/m²
* Severe hepatic insufficiency (Child-Pugh class C)
* Contraindication to NATISPRAY 0.30 mg/dose, solution for oral spray (and in particular hypersensitivity to nitrates in accordance with the SPC (Summary of Product Characteristics) of NATISPRAY)
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection, or guardianship or curatorship
* Previous or current treatment with Belatacept
* Severe high blood pressure (DBP ≥ 110 mm Hg and/or SBP ≥ 180 mm Hg)
* Presence or history of functional or ligated or thrombosed bilateral arteriovenous fistula, preventing explorations
* Pregnant, breastfeeding woman, or absence of proven effective contraception
* Excessive alcohol consumption (no more than 10 drinks per week)
* Active smoking with a daily consumption of more than 21 mg of nicotine per day or taking nicotine substitutes with a dose greater than 21 mg/24 hours
* Drug addiction or suspected illicit drug use
* Patient participating or having participated in the 4 weeks preceding inclusion in a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Replacement of anticalcineurins with Belatacept in kidney transplant patients allows an improvement in the endothelium-dependent dilation of peripheral conductance arteries | at 6 months
  The primary endpoint is to compare the variation over 6 months in the amplitude of endothelium-dependent dilation during the post-ischemic hyperemia maneuver (Paragraph 7.1) (visit V2 and V3) measured by vascular ultrasound with a automated software analysis in real time between the Bélatacept group and the anticalcineurin group.

IPD SHARING:
Plan to Share IPD: No